CLINICAL TRIAL: NCT00832975
Title: Study of Slow Ventricular Tachycardia and Atrial Fibrillation Incidence Documented by Intracardiac Electrogram in Patients Implanted With an Implantable Cardiac Device (ICD) .
Brief Title: AVAI: Atrial Ventricular Arrythmia Incidence
Acronym: AVAI
Status: Completed | Type: Observational
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Other Study IDs: CR08003ES
Record Dates: First submitted 2009-01-29; First posted 2009-01-30 (Estimated); Results first posted 2015-03-03 (Estimated); Last update posted 2019-02-21 (Actual); Status verified 2019-02

CONDITIONS: Ventricular Tachycardia; Atrial Fibrillation
MeSH Terms: conditions — Tachycardia, Ventricular; Atrial Fibrillation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this observational study is to collect data regarding the population of patients implanted with St. Jude Medical ICD.

DETAILED DESCRIPTION:
The purpose of this observational study is to collect data regarding the population of patients implanted with a St. Jude Medical ICD. Data regarding Slow Ventricular Tachycardia Episodes, Atrial Fibrillation Episodes and the devices programmed parameters will be collected during two years after the implant.

ELIGIBILITY:
Inclusion Criteria:

* Patient has been implanted with a St Jude Medical ICD, mono,bicameral or cardiac resynchronization therapy - Defibrillator (CRT-D) according the American College of Cardiology (ACC), American Heart Association (AHA), National Standards for Physical Education (NASPE) guidelines. (min. 24 hours - max. 2 months)
* Patient has signed the study specific Informed consent document.
* Patient is older than 18 years of age

Exclusion Criteria:

* Patient has a permanent Atrial Fibrillation
* Patient has a documented slow ventricular Tachycardia Episodes previous to the ICD implant.
* Patient not programed with a ventricular Tachycardia (VT) zone upper than 120 bpm.
* Patient requires cardiac resynchronization
* Patient has Brugada Syndrome
* Patient has long QT Syndrome
* Patient has a device replacement;
* Patient is pregnant or nursing
* Patient is unable to attend the follow-up visits

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients implanted with a St. Jude Medical ICD
Sampling Method: Non-Probability Sample
Enrollment: 157 (Actual)
Dates: Start 2008-12; Primary Completion 2013-02 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ignacio Fernández Lozano, PhD., Principal Investigator — Hospital Universitario Puerta de Hierro; Javier Alzueta, PhD, Principal Investigator — Hospital Clinico Universitario Virgen de la Victoria
Locations (2):
- Spain (2):
  - Hospital Universitario Puerta de Hierro, Madrid
  - Hospital Clínico Universitario Virgen de la Victoria, Málaga

RESULTS

PARTICIPANT FLOW:
Groups:
- St Jude Medical ICD/CRT-D: St Jude Medical Implantable Cardioverter Defibrillator (ICD) / Cardiac Resynchronization Therapy-Defibrillator (CRT-D) Device implanted patients
Period: Overall Study
Arm/Group | St Jude Medical ICD/CRT-D
Started | 157
Completed | 118
Not Completed | 39
Not completed — Lost to Follow-up | 7
Not completed — Protocol Violation | 6
Not completed — Death | 5
Not completed — Physician Decision | 4
Not completed — Withdrawal by Subject | 3
Not completed — Other reasons | 14

BASELINE CHARACTERISTICS:
Population: All patients
Groups:
- St Jude Medical ICD/CRT-D: St Jude Medical ICD/CRT-D Device implanted patients
Arm/Group | St Jude Medical ICD/CRT-D
Number analyzed (Participants) | 157
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.67 (13.39)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35
  Male | 122

OUTCOME MEASURES:

1. Primary Outcome: Slow Ventricular Tachycardia Episodes Devices Detected (Between 120-150 Bpm and > 30sec) Atrial Fibrillation (AF) Episodes Devices Detected (> 30 Sec)
Description: Slow Ventricular Tachycardia episodes will be considered as a tachycardia episodes detected by the device between 120-150 bpm and with more than 30sec of duration AF Episodes will be considered only when their duration is >30sec
Time Frame: 24 months
Population: 157 patients were analyzed: 118 completed 2 years of Follow Up (FU) and 39 patients were terminated before completing it
Measure: Number; unit: Episodes
Arm/Group | St Jude Medical ICD/CRT-D
Number analyzed (Participants) | 157
Episodes
  Device Slow VT Episodes | 3778
  Internal Investigator Slow VT Episodes | 112
  External investigator Slow VT Episodes | 68
  Device AF>30sec Episodes | 308
  Internal Investigator AF>30sec Episodes | 1900
  External Investigator AF>30sec Episodes | 2864

2. Secondary Outcome: Cardiovascular Mortality Hospitalization Rate Due to Cardiovascular Reasons or Heart Failure
Time Frame: 24 months
Measure: Number; unit: Patients
Arm/Group | St Jude Medical ICD/CRT-D
Number analyzed (Participants) | 157
Patients
  Cardiovascular Mortality | 5
  Hospitalization due to cardiovascular reasons | 31

ADVERSE EVENTS:
Time Frame: 2 years
Description: All Adverse Events (AE) in the study were classified as:
  * Serious AE
  * Serious Device Related AE
  * Unsuspected Serious Device Related AE
  * Non-Serious AE
  * Non-Serious Device Related AE
  There is not enough information available for a more detailed classification
Arm/Group | St Jude Medical ICD/CRT-D
Serious Adverse Events (participants affected / at risk) | 67/157
Other Adverse Events (participants affected / at risk) | 20/157
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | St Jude Medical ICD/CRT-D (N=157)
Serious AE (General disorders) | 51 (88)
Serious Device related AE (Cardiac disorders) | 13 (14)
Unspected Serious Device related AE (Cardiac disorders) | 3 (3)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | St Jude Medical ICD/CRT-D (N=157)
AE (General disorders) | 16 (19)
Device related AE (General disorders) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No